CLINICAL TRIAL: NCT04642703
Title: Mortality in Patients With Severe SARS-CoV-2 Pneumonia Who Underwent Tracheostomy Due to Prolonged Mechanical Ventilation
Brief Title: Mortality in Patients With Severe COVID-19 Pneumonia Who Underwent Tracheostomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Carlos Romero, MD., Medical Chief, Intensive Care Unit, Hospital Clínico Universidad de Chile, University of Chile
Other Study IDs: 65/20
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Ventilation; Covid19; Tracheostomy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 ventilated patients subjected to tracheostomy: Patients who receive percutaneous or surgical tracheostomy due to prolonged mechanical ventilation. The indication is made by an experts team and based on national guidelines
- COVID-19 ventilated patients without tracheostomy: Patients supported with mechanical ventilation by 10 days or more in who an experts team of physicians decided do not perform a tracheostomy

SUMMARY:
Background: Invasive mechanical ventilation (IMV) in COVID-19 patients has been associated with a high mortality rate. In this context, the utility of tracheostomy has been questioned in this group of ill patients. This study aims to compare in-hospital mortality in COVID-19 patients with and without tracheostomy due to prolonged IMV Methods: Cohort study of adult COVID-19 patients subjected to prolonged IMV. Since the first COVID-19 case (March 3, 2020) up to November 30, 2020, all adult critical patients supported with IMV by 10 days or more at the Hospital Clínico Universidad de Chile will be included in the cohort. Pregnant women and non-adult patients will be excluded. Baseline characteristics, comorbidities, laboratory data, disease severity, and ventilatory support will be retrospectively collected from clinical records. The indication of tracheostomy, as part of our standard of care, will be indicated by a team of specialists in intensive care medicine, following national guidelines, and consented to by the patient's family. The 90-days mortality rate will be the primary outcome, whereas IMV days, hospital/CU length of stay, and the frequency of healthcare-associated infections will be the secondary outcomes. Also, a follow-up interview will be performed one year after a hospital discharged in order to assess the vital status and quality of life.

The mortality of patients subjected to tracheostomy will be compared with the group of patients without tracheostomy by logistic regression models. Furthermore, propensity-score methods will be performed as a complementary analysis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 confirmed case
* Invasive mechanical ventilation by 10 days or longer

Exclusion Criteria:

* Childhood
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients with respiratory failure needing mechanical ventilation for 10 days or longer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
90-days mortality rate | Since mechanical ventilation onset to death or 90-days follow-up
  Death occurred during the follow-up

SECONDARY OUTCOMES:
Hospital length of stay | From hospital admission to discharge, up to 90 days
  Days from hospital admission to discharge
ICU length of stay | From first ICU admission to transfer at a lower complexity unit, up to 90 days
  Days elapsed in the first ICU admission
Time of mechanical ventilation | From orotracheal intubation to mechanical ventilation extubation (weaning), up to 90 days
  Days of invasive ventilatory support
Health-care associated infections | From hospital admission to discharge, up to 90 days
  Frequency of respiratory, urinary tract, blood stream and invasive device-related infections
Long-term quality of life assessed by Short Form-36 Health Survey, SF-36 | One year after hospital discharge
  Score on the the Short Form-36 Health Survey (SF-36). SF-36 is a 36-item questionary that assesses the quality of life on eight health-related aspects. It scores from 0 (maximum disability) to 100 (no disability): the lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Romero, MD, Principal Investigator — Intensive Care Unit, Hospital Clínico Universidad de Chile, University of Chile
Locations (1):
- Intensive Care Unit, Hospital Clínico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided